CLINICAL TRIAL: NCT04532957
Title: A Phase I, Double Blind, Placebo Controlled, Multiple Oral Dose, Safety, Tolerability, and Pharmacokinetic Study of KBP-7072 in Healthy Male and Female Subjects
Brief Title: A Multiple Ascending Dose Study to Investigate Safety of KBP-7072 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KBP Biosciences (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KBP7072-1-003
Record Dates: First submitted 2020-07-06; First posted 2020-08-31 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: KBP-7072; Multiple ascending dose; Healthy Subjects; Antibiotics; Tetracycline
MeSH Terms: interventions — kbp-7072

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Multiple doses 100mg Healthy subjects receive multiple doses of KBP-7072 (100mg) or Placebo (100mg) QD capsules daily for a total of 10 days
  Interventions: Drug: KBP-7072; Drug: Placebo
- Group 2 (Experimental): Multiple doses 200mg Healthy subjects receive multiple doses of KBP-7072 (200mg) or Placebo (200mg) QD capsules daily for a total of 10 days
  Interventions: Drug: KBP-7072; Drug: Placebo
- Group 3 (Experimental): Multiple doses dose tbd Healthy subjects receive multiple doses of KBP-7072 (tbd) or Placebo(tbd) QD capsules daily for a total of 10 days
  Interventions: Drug: KBP-7072; Drug: Placebo

INTERVENTIONS:
Drug: KBP-7072 — QD oral capsules
Drug: Placebo — matching placebo capsules

SUMMARY:
This is a double-blind, placebo-controlled, multiple oral dose study to evaluate safety, tolerability, and pharmacokinetic of KBP-7072 in healthy subjects.

DETAILED DESCRIPTION:
This was a double-blind, randomized, placebo-controlled, parallel-group, multiple oral dose study. Overall, a total of 24 subjects were studied in 3 groups (Groups 1 to 3); with each group consisting of 8 subjects (6 subjects receiving KBP-7072 and 2 subjects receiving placebo). Groups 1 and 2 evaluated 100 and 200 mg QD, respectively. The dose level of 150 mg QD evaluated in Group 3 was determined based on data obtained from Group 2 of this stud

ELIGIBILITY:
Inclusion Criteria:

1. Females of nonchildbearing potential or males, of any race, between 18 and 50 years of age, inclusive, at screening.
2. Body mass index between 18.0 and 30.0 kg/m2, inclusive, at screening.
3. In good health, determined by no clinically significant findings from medical history, physical and ophthalmologic examinations, 12 lead ECG, vital sign measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and check in as assessed by the investigator (or designee).
4. Females of nonchildbearing potential defined as permanently sterile or postmenopausal. Males will agree to use contraception.
5. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
3. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed). Cholecystectomy will not be allowed.
4. Alanine aminotransferase or AST ≥ 1 × ULN. Assessments may be repeated once if outside the range at screening and/or check-in, at the discretion of the investigator.
5. Fibroscan controlled attenuation parameter (CAP) > 238 dB/m and vibration controlled transient elastography (VCTE) > 7 kPa.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Safety of KBP-7072 by assessing the number and severity of adverse events, laboratory abnormalities, ECGs, vital signs, and physical examinations. | Day 1 - 10
  Safety Assessment evaluated through adverse events, laboratory evaluations, vital signs, ECGs, and physical examinations

SECONDARY OUTCOMES:
Pharmacokinetics Parameters: Area under the plasma concentration-time curve (AUC) from time zero to time of last quantifiable concentration (AUC0-tlast), | Day 1 predose and at 0.5, 1, 2, 4, 6, 10, 12, 18, and 24 hours postdose; on Days 4, 7, 8 and 9 predose and on Day 10 predose and at 0.5, 1, 2, 4, 6, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours postdose.
  Area under the plasma concentration-time curve (AUC) from time zero to time of last quantifiable concentration (AUC0-tlast) - Plasma
Pharmacokinetics Parameters: AUC over a dosing interval (AUC0-τ), from time zero to time of last quantifiable concentration (AUC0-tlast) | Day 1 predose and at 0.5, 1, 2, 4, 6, 10, 12, 18, and 24 hours postdose; on Days 4, 7, 8 and 9 predose and on Day 10 predose and at 0.5, 1, 2, 4, 6, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours postdose.
  AUC over a dosing interval (AUC0-τ) - Plamsa
Pharmacokinetics Parameters: Maximum observed plasma concentration (Cmax) | Day 1 predose and at 0.5, 1, 2, 4, 6, 10, 12, 18, and 24 hours postdose; on Days 4, 7, 8 and 9 predose and on Day 10 predose and at 0.5, 1, 2, 4, 6, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours postdose.
  Maximum observed plasma concentration (Cmax) - Plasma
Pharmacokinetics Parameters: time of the maximum observed plasma concentration (Tmax) | Day 1 predose and at 0.5, 1, 2, 4, 6, 10, 12, 18, and 24 hours postdose; on Days 4, 7, 8 and 9 predose and on Day 10 predose and at 0.5, 1, 2, 4, 6, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours postdose.
  Time of the maximum observed plasma concentration (Tmax) - Plasma
Pharmacokinetics Parameters: apparent terminal elimination half-life (t1/2) | Day 1 predose and at 0.5, 1, 2, 4, 6, 10, 12, 18, and 24 hours postdose; on Days 4, 7, 8 and 9 predose and on Day 10 predose and at 0.5, 1, 2, 4, 6, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours postdose.
  Apparent terminal elimination half-life (t1/2) - Plasma
Pharmacokinetics Parameters: observed accumulation ratio based on AUC0-τ (ARAUC0-τ) | Day 1 predose and at 0.5, 1, 2, 4, 6, 10, 12, 18, and 24 hours postdose; on Days 4, 7, 8 and 9 predose and on Day 10 predose and at 0.5, 1, 2, 4, 6, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours postdose.
  Observed accumulation ratio based on AUC0-τ (ARAUC0-τ) - Plasma
Pharmacokinetics Parameters: amount of drug excreted in urine (Ae) | Day 1 at predose (spot collection), 0-6, 6-12, and 12-24 hours postdose, on Days 4, 7, 8 and 9 at predose (spot collection) and on Day 10 at 0-6, 6-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, and 144-168 hours postdose.
  Amount of drug excreted in urine (Ae) - Urine

CONTACTS AND LOCATIONS:
Overall Officials: James McCabe, MD, Study Director — KBP Biosciences
Locations (1):
- Covance Clinical Research Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No